CLINICAL TRIAL: NCT05167539
Title: Aortic Root Enlargement Versus Aortic Root Replacement in the Management of Cases With Small Aortic Root
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Abdelraouf, Assistant Lecturer, Assiut University
Other Study IDs: Aortic valve surgery
Record Dates: First submitted 2021-12-20; First posted 2021-12-22 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Aortic Valve Disease
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mechanical aortic valve replacement: simple procedure but need long term of anticoagulant
  Interventions: Procedure: Aortic valve surgery
- Aortic root replacement: complicated procedure but without anticoagulant
  Interventions: Procedure: Aortic valve surgery

INTERVENTIONS:
Procedure: Aortic valve surgery — mechanical aortic valve replacement versus ross procedure and stentless bioprothesis

SUMMARY:
Each type of Aortic valve surgery has its advantages and disadvantages; we aim to differentiate between two types of aortic valve surgery: aortic root replacement (using either Ross procedure or stentless bioprosthesis procedure) and mechanical aortic valve replacement.

DETAILED DESCRIPTION:
Aortic valve replacement has been performed since the 1950s. Since then, the surgical procedure has been optimized to reduce the risk of procedure-related complications. In addition, technical advances in the design of valves have significantly improved long-term prognosis. After the initial use of mechanical ball-caged valves, numerous monoleaflet and bileaflet valves have been introduced and evaluated. Moreover, bioprosthetic valves came on the market in the 1960s as an alternative to mechanical valve.

The pulmonary autograft was introduced in clinical practice as a substitute for the diseased aortic valve by Donald Ross in 1967. The original implant technique, namely subcoronary freehand grafting, was associated with substantial prevalence of early and late valve dysfunction, thereby limiting widespread adoption of the operation. More recent experience with pulmonary autografts used for complete or partial aortic root replacement allowed for satisfactory functional behavior of the valve .

Homografts for aortic valve replacement were the first biologic stentless prostheses used in clinical practice in the 1960s. Binet introduced a stentless porcine bioprosthesis, but the valve was abandoned because of poor tissue fixation. Due to limited availability and a relatively difficult implantation technique, mechanical AVR became the popular therapeutic option. The disadvantage of life-long anticoagulation therapy in mechanical AVR prompted the development of xenogeneic bioprostheses. Although porcine aortic valves or pericardial tissue mounted on a stent made the implantation technique easier, these valves sacrificed orifice area and increased stress at the attachment of the stent, which caused earlier primary tissue failure. Optimizing hemodynamics to prevent patient-prosthetic mismatch and improve durability revived the use of stentless bioprostheses in the early 1990s.

Patients with an expected survival of less than 10 years (more than 65 years old, renal disease, lung disease, patients who are more than 60 years old), ejection fraction of less than 40%, or coronary disease would be reasonable candidates for aortic bioprostheses to avoid anticoagulation with an extremely low likelihood of aortic valve reoperation. Results tend to favor mechanical aortic valves in patients under age 65 years with a life expectancy of at least 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing Aortic valve surgery.

Exclusion Criteria:

* Patients who have other procedure with aortic valve surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who presented to Cardiothoracic Surgery Department, Assiut University Heart Hospital and Aswan heart center who meet the listed inclusion will be eligible for the study. The charts will be reviewed and eligible patients will be filtered
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-02-10 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with failure of surgery | baseline
  Number of participants with failure of initial intervention , Requiring a second intervention i.e redo aortic valve surgery